CLINICAL TRIAL: NCT00853489
Title: RhBMP-2 vs. Autograft for Critical Size Tibial Defects: A Multicenter Randomized Trial
Brief Title: rhBMP-2 Versus Autograft in Critical Size Tibial Defects
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment too slow
Sponsor: St. Louis University (Other)
Collaborators: Major Extremity Trauma Research Consortium (Other)
Responsible Party: Principal Investigator, Thomas Revak, DO, Instructor, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: W81XWH-09-20108; 15915 (Other: Saint Louis University Institutional Review Board)
Record Dates: First submitted 2009-02-24; First posted 2009-03-02 (Estimated); Results first posted 2018-03-13 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Tibial Fractures
Keywords: Open tibia fractures; rhBMP-2; critical size defects; bone grafting
MeSH Terms: conditions — Tibial Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- recombinant bone morphogenetic protein 2 (Experimental): The patient will receive rhBMP-2 plus allograft chips in the bone defect site. Intervention type: surgical
  Interventions: Device: recombinant bone morphogenetic protein 2
- Autogenous iliac crest bone graft (Active Comparator): Bone will be harvested from the iliac crest and placed in the bone defect.
  Interventions: Procedure: Autogenous iliac crest bone graft

INTERVENTIONS:
Device: recombinant bone morphogenetic protein 2 — Patients will receive 1.50 mg/ml -12 mg of rhBMP-2 soaked on a absorbable collagen sponge (rhBMP-2/ACS) as an adjuvant to a freeze-dried cancellous allograft
  Other Names: (rhBMP-2) (INFUSE)
  Arms: recombinant bone morphogenetic protein 2
Procedure: Autogenous iliac crest bone graft — Patients will undergo autogenous iliac crest bone graft surgery per the surgeon's usual practice.
  Arms: Autogenous iliac crest bone graft

SUMMARY:
The purpose of our study is to evaluate the use of recombinant human bone morphogenetic protein 2 (RhBMP-2) as compared to standard ICBG in the treatment of severe open tibia fractures with a critical size bone defect (at least one centimeter in length compromising at least 50% of the circumference of the bone).

DETAILED DESCRIPTION:
Open tibia fractures have a 15% or higher rate of not healing. Those fractures which do not heal are typically treated with bone from the hip (iliac crest autograft; or ICBG). The use of ICBG bone with the treatment of delayed unions/non-unions with critical defect, although successful, has its drawbacks. The bone graft sources are limited and the procedure is associated with additional operating room time plus a second incision with increased risk of infection, post operative pain and increased hospital stay. The purpose of this study is to determine if Rh-BMP2, a new bone graft substitute, is at least as effective as using bone from the hip (autograft) to help promote healing of open, tibia (shin bone) fractures.

Research Questions:

Primary:

What is the relative effect of rhBMP-2 versus autogenous ICBG on rates of union in patients with critical size defects following tibial shaft fractures?

Null hypothesis #1: rhBMP-2 has the same union rate when used in critical-sized defects as does ICBG.

Secondary:

What is the relative effect of rhBMP-2 versus autogenous ICBG on infection rates in patients with nonunion or critical size defects following tibial shaft fractures?

Null hypothesis #2: The infection rate in open tibias with critical-sized defects treated with rhBMP-2 and autogenous ICBG are the same.

What is the economic impact of the use of Rh-BMP 2 for tibial fractures with critical sized defects?

Null hypothesis #3: There will be no difference in the economic cost of the treatment of critical sized defects using the RhBMP-2 versus iliac crest bone graft.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-65 years old with an open tibia fracture involving diaphysis (if patient has a bilateral tibia fracture and both require a bone graft, then each will be randomized separately).
* Tibia fractures with a circumferential bone defect of at least one centimeter in length compromising at least 50% of the circumference of the bone.
* The definitive treatment of the tibia fracture must be with an intramedullary nail (may have temporary external fixation prior to IM nail placement).
* Patients whose treatment plan includes placement of a bone graft between 6 to 16 weeks after their initial injury.
* Patients who have no evidence of infection by clinical examination (defined as active infection at the operative site, purulent drainage from the fracture or evidence of active osteomyelitis at the time of bone graft).
* Patients who are independent in living and ambulation prior to injury.
* Patients who are English speaking.
* Patients who are willing to provide consent and available for follow-up for at least 12 months following definitive surgical procedure.

Exclusion Criteria:

* Patients who are pregnant or lactating.
* Patients with known hypersensitivity to rhBMP-2 or bovine type I collagen.
* Patients with a history of tumor, a resected or extant tumor, an active malignancy, or patients undergoing treatment for malignancy.
* Patients who are skeletally immature (<18 years of age or no radiographic evidence of epiphyseal closure).
* Patients with inadequate neurovascular status, e.g. high risk of amputation.
* Patients with compartment syndrome of the affected limb.
* Patients with immune deficiency or history of auto-immune disease,
* Patients who have undergone treatment of any other investigational therapy within the month preceding implantation or planned within the 12 months following implantation.
* Patients unable to return for required follow-up visits.
* Patients who have medical co-morbidities that preclude treatment with a general anesthetic.
* Patient who is pending incarceration or who is incarcerated.
* Patients with an active infection at the operative site, purulent drainage from the fracture or evidence of active osteomyelitis at the time of bone grafting.
* Patient has intraoperative positive gram stain or an elevated CRP after laboratory screening for infection.
* Patient has segmental defects longer than 5cm in length.
* Patients who have segmental defects that require more than 60 cc of bone graft.
* Patients who require more than one large kit of rhBMP-2 at time of surgery.
* Patient's anticipated treatment plan also includes the use of other procedures to promote fracture healing, e.g. ultrasound, magnetic field or electrical stimulation.
* Patient's tibia fracture has been treated with additional fixation beyond the intramedullary nail, e.g. plates, wires or screws.
* Patients who have pathological fractures; a known history of Paget's disease or known history of heterotropic calcification.
* Patients with a Glasgow Coma Scale less than 15 (less than fully awake) at the time of informed consent.
* Patients with previous hardware in place that prevents placement of an intramedullary nail for treatment of the tibial shaft fracture.
* Patients with prior use of INFUSE.

If the patient is a female of child bearing potential:

* Does she have a negative pregnancy test (administered within 72 hours prior to surgery)?
* Has she agreed to use adequate contraception for a period of at least 1 year following implementation of rhBMP-2?

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-08; Primary Completion 2017-02-17 (Actual); Study Completion 2017-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Revak, DO, Principal Investigator — St. Louis Medical Center; Paul Tornetta, MD, Principal Investigator — Boston Medical Center
Locations (13):
- United States (13):
  - UCSF Medical Center, San Francisco, California
  - Denver Health and Hospital Authority, Denver, Colorado
  - Florida Orthopaedic Institute / Tampa General & St. Joseph's Hospitals, Tampa, Florida
  - University of Iowa Hospitals, Iowa City, Iowa
  - Boston Medical Center, Boston, Massachusetts
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - St. Louis Medical Center, St Louis, Missouri
  - Carolinas Medical Center, Charlotte, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - University of Oklahoma / OU Medical Center, Oklahoma City, Oklahoma
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Washington / Harborview Medical Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 34 consented One was inelgible at time of graft due to infection pre enrollment Two were outside study period One Administrative withdrawl Total randomized : 30
Period: Overall Study
Arm/Group | Recombinant Bone Morphogenetic Protein 2 | Autogenous Iliac Crest Bone Graft
Started | 16 | 14
Completed | 11 | 12
Not Completed | 5 | 2
Not completed — Lost to Follow-up | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Recombinant Bone Morphogenetic Protein 2 | Autogenous Iliac Crest Bone Graft | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 14 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (12) | 35 (12) | 36 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 12 | 11 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 14 | 11 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 13 | 13 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 14 | 30
Count of participants [Count of Participants; unit: Participants] | 16 | 14 | 30

OUTCOME MEASURES:

1. Primary Outcome: Fracture Healing (Union) at 12 Months
Description: Union will be defined by:
  1. Radiographic union as defined by the Radiographic union scale in tibia fractures (RUST) score, Radiographic evaluation will be assessed by blinded orthopaedic surgeons.
Time Frame: 12 months post op
Population: RUST scores were used to determine radiograpghic union at 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Recombinant Bone Morphogenetic Protein 2 | Autogenous Iliac Crest Bone Graft
Number analyzed (Participants) | 12 | 11
Participants | 12 | 11

2. Secondary Outcome: Infection
Description: Infection will be assessed based on the CDC criteria for deep and superficial infection.
Time Frame: 12 months post op.
Population: Infection was decribed in protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Recombinant Bone Morphogenetic Protein 2 | Autogenous Iliac Crest Bone Graft
Number analyzed (Participants) | 16 | 14
Participants | 3 | 0

3. Secondary Outcome: Medical Cost
Description: An economic evaluation will also be performed including the costs of iliac crest bone graft harvest and complications from the bone graft surgery and the cost of the Rh-BMP 2 and the biologic implant used in the treatment group.
Time Frame: 12 mos post op
Population: Hospital bills for bone graft surgery admission were available on 25 patients total
Measure: Mean (Full Range); unit: dollars for total admission cost
Arm/Group | Recombinant Bone Morphogenetic Protein 2 | Autogenous Iliac Crest Bone Graft
Number analyzed (Participants) | 12 | 13
dollars for total admission cost | 13033 [9038 to 22041] | 7535 [2480 to 22915]

ADVERSE EVENTS:
Time Frame: One year after enrollment
Description: The definition of adverse events/SAE does not differ from clinicaltrials.gov
Arm/Group | Recombinant Bone Morphogenetic Protein 2 | Autogenous Iliac Crest Bone Graft
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/14
Serious Adverse Events (participants affected / at risk) | 3/16 | 0/14
Other Adverse Events (participants affected / at risk) | 1/16 | 1/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recombinant Bone Morphogenetic Protein 2 (N=16) | Autogenous Iliac Crest Bone Graft (N=14)
Infection (Surgical and medical procedures) | 3 (3) | 0 (0) — Infection definition described in protocol
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recombinant Bone Morphogenetic Protein 2 (N=16) | Autogenous Iliac Crest Bone Graft (N=14)
Non union (Surgical and medical procedures) | 1 (1) | 1 (1) — Defined in protocol

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-01-02): https://cdn.clinicaltrials.gov/large-docs/89/NCT00853489/Prot_SAP_000.pdf